CLINICAL TRIAL: NCT01242111
Title: A Multicenter, Multinational, Open-Label, Extension Study to Evaluate the Long-Term Efficacy and Safety of BMN 110 in Patients With Mucopolysaccharidosis IVA (Morquio A Syndrome)
Brief Title: A Study to Evaluate the Long-Term Efficacy and Safety of BMN 110 in Patients With Mucopolysaccharidosis IVA (Morquio A Syndrome)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOR-100
Record Dates: First submitted 2010-10-28; First posted 2010-11-16 (Estimated); Results first posted 2015-09-30 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-08

CONDITIONS: MPS IV A; Mucopolysaccharidosis IVA; Morquio A Syndrome
Keywords: Mucopolysaccharidosis IV type A; MPS IV Type A; Mucopolysaccharidosis IVA; MPS IVA; Morquio A Syndrome; Lysosomal Storage Disorder; LSD; N-acetylgalactosamine-6-sulfatase; N-acetylgalactosamine-6-sulfate sulfatase; galactose-6-sulfatase; GALNS; enzyme replacement therapy; ERT
MeSH Terms: conditions — Mucopolysaccharidosis IV; Lysosomal Storage Diseases | interventions — GALNS protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMN 110 (Experimental)
  Interventions: Drug: BMN 110

INTERVENTIONS:
Drug: BMN 110 — Patients will receive an intravenous infusion of BMN110 at 2.0mg/kg/week, over a period of approximately 4 hours per infusion, for up to 240 weeks.

SUMMARY:
This multicenter, open-label extension study is designed to assess long-term efficacy and safety of 2.0 milligrams (mg)/kilogram(kg)/week of BMN 110 in patients diagnosed with Mucopolysaccharidosis IVA (MPS IVA). Patients with MPS IVA, who enrolled in a prior BioMarin sponsored clinical study of BMN 110 (NCT00884949; Study Identification Number MOR-002), were eligible to enroll in this study (except patients who enrolled in NCT01275066; Study Identification Number MOR-004).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written, signed informed consent, or in the case of patients under the age of 18 (or 16 years, depending on the region), provide written assent (if required) and written informed consent by a legally authorized representative after the nature of the study has been explained, and prior to any research-related procedures.
* Sexually active patients must be willing to use an acceptable method of contraception while participating in the study.
* Females of childbearing potential must have a negative pregnancy test at Baseline and be willing to have additional pregnancy tests during the study.
* Must have enrolled in a prior BioMarin sponsored clinical study of BMN 110.

Exclusion Criteria:

* Pregnant or breastfeeding at Baseline or planning to become pregnant (self or partner) at any time during the study.
* Use of any investigational product (other than BMN 110 in a prior clinical study) or investigational medical device within 30 days prior to Baseline, or requirement for any investigational agent prior to completion of all scheduled study assessments.
* Concurrent disease or condition, including but not limited to symptomatic cervical spine instability, clinically significant spinal cord compression, or severe cardiac disease that would interfere with study participation or safety as determined by the Investigator.
* Any condition that, in the view of the Investigator, places the patient at high risk of poor treatment compliance or of not completing the study.
* Were enrolled in MOR-004 (patients from MOR-004 may be eligible to participate in a separate, appropriately designed, extension study).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Decker, MD, Study Director — BioMarin Pharmaceutical
Locations (4):
- United Kingdom (4):
  - Birmingham, United Kingdom
  - Dumfries, United Kingdom
  - London, United Kingdom
  - Manchester, United Kingdom

REFERENCES:
- [Derived] Hendriksz C, Santra S, Jones SA, Geberhiwot T, Jesaitis L, Long B, Qi Y, Hawley SM, Decker C. Safety, immunogenicity, and clinical outcomes in patients with Morquio A syndrome participating in 2 sequential open-label studies of elosulfase alfa enzyme replacement therapy (MOR-002/MOR-100), representing 5 years of treatment. Mol Genet Metab. 2018 Apr;123(4):479-487. doi: 10.1016/j.ymgme.2018.02.011. Epub 2018 Feb 19. PMID 29526614
- See also: BioMarin Pharmaceutical Inc. website — http://www.bmrn.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BMN 110
Started | 20
Completed | 17
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Did not consent to MOR-100 follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | BMN 110
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.4 (2.90)
Age, Customized [Number; unit: participants]
  >=4 to < 8 years | 10
  >=8 to <10 years | 5
  >=10 to <=18 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  Other | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20

OUTCOME MEASURES:

1. Primary Outcome: Safety Evaluation
Description: The primary objective of the study is to evaluate the safety of weekly infusions of BMN 110; the safety variables included Adverse Events (AEs).
  The primary outcome measure data is presented in more detail under the Adverse Events section.
Time Frame: Entire Study Period, up to 240 weeks
Population: The primary outcome measure data is presented in more detail under the Adverse Events section.
Measure: Number; unit: participants
Arm/Group | BMN 110
Number analyzed (Participants) | 20
participants
  Serious Adverse Events | 19
  Other (Not Including Serious) Adverse Events | 20

2. Secondary Outcome: Change From Baseline in Endurance as Measured by the 6-minute Walk Test During the Pilot Trial (MOR-002) and Current Extension Trial (MOR-100).
Description: Change from baseline in meters in 6-minute Walk Test. As a measure of endurance, a 6-minute walk test (6MWT) was performed according to the American Thoracic Society Guidelines. Patients were instructed to walk as far as possible in 6 minutes.
Time Frame: Baseline and every 12 weeks for up to 72 weeks during the MOR-002 pilot trial and every 24 weeks for up to 192 weeks during the MOR-100 extension trial
Population: Intent-to-Treat population (all subjects who enrolled in the study). Two patients were either physically (score was designated as 0 m) or developmentally (score was set to missing) unable to perform the 6MWT. The analysis was based on observed cases.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | BMN 110
Number analyzed (Participants) | 20
meters
  MOR-002 Week 12 Change from Baseline (n=19) | -20.7 (85.95)
  MOR-002 Week 24 Change from Baseline (n=17) | 16.3 (71.74)
  MOR-002 Week 36 Change from Baseline (n=17) | 13.8 (63.25)
  MOR-002 Week 48 Change from Baseline (n=17) | -4.8 (64.70)
  MOR-002 Week 72 Change from Baseline (n=17) | 4.0 (87.24)
  MOR-100 Week 0 Change from Baseline (n=16) | 15.7 (89.00)
  MOR-100 Week 24 Change from Baseline (n=16) | 24.5 (101.23)
  MOR-100 Week 48 Change from Baseline (n=16) | 6.8 (98.66)
  MOR-100 Week 72 Change from Baseline (n=17) | -49.8 (132.63)
  MOR-100 Week 96 Change from Baseline (n=16) | 11.2 (85.24)
  MOR-100 Week 120 Change from Baseline (n=16) | 4.2 (94.09)
  MOR-100 Week 144 Change from Baseline (n=13) | 3.1 (106.82)
  MOR-100 Week 192 Change from Baseline (n=9) | -37.1 (103.96)

3. Secondary Outcome: Change in Baseline in Endurance as Measured by the 3 Minute Stair Climb During the Pilot Trial (MOR-002) and Current Extension Trial (MOR-100).
Description: Change from baseline in the 3-minute Stair Climb Test (3MSCT). Patients walked up stairs that have a railing, which could be used for support, for 3 minutes, with the number of stairs climbed recorded. The test result was the number of steps climbed per minute.
Time Frame: as for outcome 2
Population: Intent-to-Treat population (all subjects who enrolled in the study). One patient was developmentally unable to perform the 3MSCT and the test scores were set to missing. The analysis was based on observed cases.
Measure: Mean (Standard Deviation); unit: steps/min
Arm/Group | BMN 110
Number analyzed (Participants) | 20
steps/min
  MOR-002 Week 12 Change from Baseline (n=19) | 0.3 (14.07)
  MOR-002 Week 24 Change from Baseline (n=17) | 6.1 (8.66)
  MOR-002 Week 36 Change from Baseline (n=17) | 7.8 (13.69)
  MOR-002 Week 48 Change from Baseline (n=17) | 9.7 (14.42)
  MOR-002 Week 72 Change from Baseline (n=17) | 9.7 (13.91)
  MOR-100 Week 0 Change from Baseline (n=16) | 12.7 (13.96)
  MOR-100 Week 24 Change from Baseline (n=16) | 13.4 (17.07)
  MOR-100 Week 48 Change from Baseline (n=16) | 6.6 (16.87)
  MOR-100 Week 72 Change from Baseline (n=16) | -1.4 (21.11)
  MOR-100 Week 96 Change from Baseline (n=16) | 9.9 (18.84)
  MOR-100 Week 120 Change from Baseline (n=16) | 6.2 (14.41)
  MOR-100 Week 144 Change from Baseline (n=12) | 5.4 (11.93)
  MOR-100 Week 192 Change from Baseline (n=7) | -0.2 (10.34)

4. Secondary Outcome: Percent Change From Baseline in Urine Keratan Sulfate (uKS) Levels During the Pilot Trial (MOR-002) and Current Extension Trial (MOR-100).
Description: Percent Change from baseline in Normalized Urine KS. The percent change was calculated (Week X value - baseline value)/baseline value *100%
Time Frame: Baseline and every 12 weeks for up to 72 weeks during the MOR-002 pilot trial and every 24 weeks for up to 168 weeks during the MOR-100 extension trial
Population: Intent-to-Treat population (all subjects who enrolled in the study). The analysis was based on observed cases.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | BMN 110
Number analyzed (Participants) | 20
percentage change
  MOR-002 Wk 12 Percent Change from Baseline (n=19) | -23.2 (19.04)
  MOR-002 Wk 24 Percent Change from Baseline (n=18) | -27.9 (17.92)
  MOR-002 Wk 36 Percent Change from Baseline (n=18) | -40.6 (20.16)
  MOR-002 Wk 72 Percent Change from Baseline (n=17) | -32.2 (17.10)
  MOR-100 Wk 0 Percent Change from Baseline (n=17) | -30.0 (19.23)
  MOR-100 Wk 24 Percent Change from Baseline (n=17) | -43.6 (19.56)
  MOR-100 Wk 48 Percent Change from Baseline (n=16) | -41.9 (19.29)
  MOR-100 Wk 72 Percent Change from Baseline (n=12) | -36.4 (36.70)
  MOR-100 Wk 96 Percent Change from Baseline (n=17) | -49.7 (19.93)
  MOR-100 Wk 120 Percent Change from Baseline (n=16) | -49.3 (22.28)
  MOR-100 Wk 144 Percent Change from Baseline (n=16) | -56.6 (19.54)
  MOR-100 Wk 168 Percent Change from Baseline (n=15) | -58.9 (16.02)

5. Secondary Outcome: Percent Change From Baseline in Respiratory Function Test MVV During the Pilot Trial (MOR-002) and Current Extension Trial (MOR-100).
Description: Percent Change from baseline in Maximum Voluntary Ventilation.
Time Frame: as for outcome 2
Population: Intent-to-Treat population (all subjects who enrolled in the study). The analysis was based on observed cases.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | BMN 110
Number analyzed (Participants) | 20
percentage change
  MOR-002 Wk 12 Percent Change from Baseline (n=14) | 9.9 (21.29)
  MOR-002 Wk 24 Percent Change from Baseline (n=13) | 11.0 (21.48)
  MOR-002 Wk 36 Percent Change from Baseline (n=14) | 10.5 (17.43)
  MOR-002 Wk 72 Percent Change from Baseline (n=14) | 18.4 (20.77)
  MOR-100 Wk 0 Percent Change from Baseline (n=13) | 11.1 (16.44)
  MOR-100 Wk 24 Percent Change from Baseline (n=13) | 9.8 (22.25)
  MOR-100 Wk 48 Percent Change from Baseline (n=12) | 3.5 (17.78)
  MOR-100 Wk 72 Percent Change from Baseline (n=13) | 10.1 (27.83)
  MOR-100 Wk 96 Percent Change from Baseline (n=12) | -4.9 (35.53)
  MOR-100 Wk 120 Percent Change from Baseline (n=13) | -3.3 (28.35)
  MOR-100 Wk 144 Percent Change from Baseline (n=11) | -3.5 (34.61)
  MOR-100 Wk 192 Percent Change from Baseline (n=6) | 28.2 (38.78)

6. Secondary Outcome: Percent Change From Baseline in Respiratory Function Test FVC During the Pilot Trial (MOR-002) and Current Extension Trial (MOR-100).
Description: Percent Change from baseline in Forced Vital Capacity.
Time Frame: as for outcome 2
Population: Intent-to-Treat population (all subjects who enrolled in the study). The analysis was based on observed cases.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | BMN 110
Number analyzed (Participants) | 20
percentage change
  MOR-002 Wk 12 Percent Change from Baseline (n=18) | 3.4 (10.85)
  MOR-002 Wk 24 Percent Change from Baseline (n=16) | 0.2 (16.60)
  MOR-002 Wk 36 Percent Change from Baseline (n=16) | 10.7 (20.81)
  MOR-002 Wk 72 Percent Change from Baseline (n=16) | 12.5 (14.88)
  MOR-100 Wk 0 Percent Change from Baseline (n=15) | 11.8 (14.97)
  MOR-100 Wk 24 Percent Change from Baseline (n=14) | 15.3 (16.31)
  MOR-100 Wk 48 Percent Change from Baseline (n=13) | 15.8 (16.56)
  MOR-100 Wk 72 Percent Change from Baseline (n=15) | 16.1 (21.96)
  MOR-100 Wk 96 Percent Change from Baseline (n=14) | 14.8 (17.36)
  MOR-100 Wk 120 Percent Change from Baseline (n=16) | 22.8 (21.14)
  MOR-100 Wk 144 Percent Change from Baseline (n=12) | 17.5 (24.32)
  MOR-100 Wk 192 Percent Change from Baseline (n=7) | 18.6 (30.98)

ADVERSE EVENTS:
Time Frame: Study Period, up to 240 weeks
Arm/Group | BMN 110
Serious Adverse Events (participants affected / at risk) | 19/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 110 (N=20)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Infusion site inflammation (General disorders) | 1 (1)
Infusion site reaction (General disorders) | 2 (3)
Malaise (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Type I hypersensitivity (Immune system disorders) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 2 (2)
Infusion site infection (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (5)
Otitis media (Infections and infestations) | 3 (3)
Pneumonia (Infections and infestations) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (3)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1)
Knee deformity (Musculoskeletal and connective tissue disorders) | 6 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Cervical cord compression (Nervous system disorders) | 2 (2)
Panic attack (Psychiatric disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Abscess drainage (Surgical and medical procedures) | 1 (2)
Bone operation (Surgical and medical procedures) | 1 (1)
Central venous catheterisation (Surgical and medical procedures) | 2 (2)
Knee operation (Surgical and medical procedures) | 2 (2)
Medical device implantation (Surgical and medical procedures) | 2 (2)
Medical device removal (Surgical and medical procedures) | 2 (2)
Orthopaedic procedure (Surgical and medical procedures) | 3 (3)
Flushing (Vascular disorders) | 1 (2)
Hypertension (Vascular disorders) | 1 (1)
Jugular vein distension (Vascular disorders) | 1 (1)
Poor venous access (Vascular disorders) | 8 (9)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 110 (N=20)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 4 (5)
Aortic valve incompetence (Cardiac disorders) | 3 (3)
Diastolic dysfunction (Cardiac disorders) | 1 (1)
Mitral valve disease (Cardiac disorders) | 2 (2)
Mitral valve incompetence (Cardiac disorders) | 3 (3)
Pulmonary valve incompetence (Cardiac disorders) | 3 (3)
Tachycardia (Cardiac disorders) | 3 (6)
Tricuspid valve incompetence (Cardiac disorders) | 3 (3)
Congenital heart valve disorder (Congenital, familial and genetic disorders) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 3 (3)
Deafness (Ear and labyrinth disorders) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (2)
Ear canal erythema (Ear and labyrinth disorders) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 1 (1)
Ear disorder (Ear and labyrinth disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 12 (41)
Ear pruritus (Ear and labyrinth disorders) | 1 (1)
Hyperacusis (Ear and labyrinth disorders) | 1 (2)
Hypoacusis (Ear and labyrinth disorders) | 2 (4)
Middle ear disorder (Ear and labyrinth disorders) | 1 (1)
Motion sickness (Ear and labyrinth disorders) | 4 (9)
Otorrhoea (Ear and labyrinth disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Tympanic membrane disorder (Ear and labyrinth disorders) | 3 (3)
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 2 (2)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 1 (2)
Conjunctivitis (Eye disorders) | 3 (4)
Dry eye (Eye disorders) | 1 (1)
Eye discharge (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1)
Eye swelling (Eye disorders) | 2 (3)
Eyelid cyst (Eye disorders) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 12 (27)
Abdominal pain upper (Gastrointestinal disorders) | 11 (33)
Constipation (Gastrointestinal disorders) | 5 (5)
Dental caries (Gastrointestinal disorders) | 3 (5)
Dental plaque (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 12 (28)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 1 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (3)
Gingival hyperpigmentation (Gastrointestinal disorders) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Lip disorder (Gastrointestinal disorders) | 1 (1)
Lip pain (Gastrointestinal disorders) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (8)
Retching (Gastrointestinal disorders) | 2 (3)
Tongue discolouration (Gastrointestinal disorders) | 1 (1)
Tooth deposit (Gastrointestinal disorders) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 5 (8)
Vomiting (Gastrointestinal disorders) | 16 (92)
Application site reaction (General disorders) | 1 (1)
Application site vesicles (General disorders) | 1 (1)
Catheter site erythema (General disorders) | 3 (9)
Catheter site extravasation (General disorders) | 7 (12)
Catheter site inflammation (General disorders) | 1 (1)
Catheter site oedema (General disorders) | 1 (1)
Catheter site pain (General disorders) | 4 (5)
Catheter site rash (General disorders) | 1 (1)
Catheter site related reaction (General disorders) | 2 (3)
Catheter site scab (General disorders) | 1 (1)
Catheter site swelling (General disorders) | 2 (6)
Chest pain (General disorders) | 1 (2)
Chills (General disorders) | 1 (1)
Device connection issue (General disorders) | 1 (1)
Device dislocation (General disorders) | 1 (2)
Device expulsion (General disorders) | 1 (2)
Device leakage (General disorders) | 1 (1)
Device malfunction (General disorders) | 1 (1)
Device occlusion (General disorders) | 3 (3)
Extravasation (General disorders) | 2 (3)
Fatigue (General disorders) | 7 (11)
Feeling hot (General disorders) | 2 (2)
Gait disturbance (General disorders) | 3 (4)
Influenza like illness (General disorders) | 3 (3)
Infusion site erythema (General disorders) | 1 (1)
Infusion site extravasation (General disorders) | 1 (2)
Infusion site pain (General disorders) | 1 (1)
Infusion site reaction (General disorders) | 1 (3)
Injection site reaction (General disorders) | 1 (1)
Local swelling (General disorders) | 2 (3)
Malaise (General disorders) | 4 (8)
Medical device complication (General disorders) | 2 (4)
Medical device site reaction (General disorders) | 1 (1)
Pain (General disorders) | 6 (12)
Pyrexia (General disorders) | 18 (103)
Vaccination site pain (General disorders) | 2 (2)
Hepatomegaly (Hepatobiliary disorders) | 1 (2)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 5 (8)
Abdominal abscess (Infections and infestations) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 6 (15)
Eye infection (Infections and infestations) | 2 (2)
Fungal infection (Infections and infestations) | 1 (1)
Fungal skin infection (Infections and infestations) | 2 (2)
Furuncle (Infections and infestations) | 3 (4)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Gingivitis (Infections and infestations) | 2 (2)
Helminthic infection (Infections and infestations) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (2)
Herpes zoster (Infections and infestations) | 2 (2)
Impetigo (Infections and infestations) | 1 (3)
Infection (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 1 (1)
Lice infestation (Infections and infestations) | 1 (2)
Localised infection (Infections and infestations) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 5 (13)
Molluscum contagiosum (Infections and infestations) | 1 (2)
Nail infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 17 (53)
Oral candidiasis (Infections and infestations) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 3 (3)
Paronychia (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 5 (8)
Skin infection (Infections and infestations) | 3 (3)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Tinea pedis (Infections and infestations) | 4 (4)
Tonsillitis (Infections and infestations) | 3 (5)
Upper respiratory tract infection (Infections and infestations) | 5 (5)
Urinary tract infection (Infections and infestations) | 1 (2)
Varicella (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 4 (5)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 6 (8)
Ear injury (Injury, poisoning and procedural complications) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 4 (4)
Eye contusion (Injury, poisoning and procedural complications) | 3 (3)
Face injury (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 8 (20)
Head injury (Injury, poisoning and procedural complications) | 8 (14)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 3 (4)
Lip injury (Injury, poisoning and procedural complications) | 1 (1)
Neck injury (Injury, poisoning and procedural complications) | 1 (1)
Occupational exposure to radiation (Injury, poisoning and procedural complications) | 1 (1)
Periorbital contusion (Injury, poisoning and procedural complications) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Procedural headache (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 7 (7)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1)
Scar (Injury, poisoning and procedural complications) | 3 (3)
Scratch (Injury, poisoning and procedural complications) | 1 (1)
Skeletal injury (Injury, poisoning and procedural complications) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Aspiration joint (Investigations) | 1 (1)
Blood cholesterol increased (Investigations) | 2 (2)
Blood immunoglobulin E increased (Investigations) | 6 (6)
Blood immunoglobulin G decreased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Blood pressure systolic increased (Investigations) | 1 (1)
Blood sodium increased (Investigations) | 1 (1)
Body temperature increased (Investigations) | 4 (6)
Breath sounds abnormal (Investigations) | 1 (1)
Cardiac murmur (Investigations) | 2 (3)
Computerised tomogram (Investigations) | 1 (1)
Electrocardiogram T wave amplitude decreased (Investigations) | 1 (2)
Eosinophil count increased (Investigations) | 2 (3)
Eosinophil percentage increased (Investigations) | 1 (1)
Liver palpable subcostal (Investigations) | 1 (1)
Nuclear magnetic resonance imaging (Investigations) | 6 (8)
Nuclear magnetic resonance imaging spinal (Investigations) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (3)
Protein total abnormal (Investigations) | 1 (1)
Protein urine (Investigations) | 1 (2)
Respiratory rate increased (Investigations) | 3 (3)
Ultrasound scan abnormal (Investigations) | 1 (1)
Weight increased (Investigations) | 2 (4)
Appetite disorder (Metabolism and nutrition disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (2)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (58)
Atlantoaxial instability (Musculoskeletal and connective tissue disorders) | 1 (1)
Axillary mass (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (17)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint instability (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2)
Knee deformity (Musculoskeletal and connective tissue disorders) | 2 (2)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 5 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 8 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 (76)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Ageusia (Nervous system disorders) | 1 (1)
Areflexia (Nervous system disorders) | 1 (1)
Cervical cord compression (Nervous system disorders) | 1 (1)
Clonus (Nervous system disorders) | 3 (4)
Dizziness (Nervous system disorders) | 4 (7)
Headache (Nervous system disorders) | 16 (100)
Lethargy (Nervous system disorders) | 5 (5)
Migraine (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Reflexes abnormal (Nervous system disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (3)
Dysuria (Renal and urinary disorders) | 1 (1)
Enuresis (Renal and urinary disorders) | 1 (3)
Incontinence (Renal and urinary disorders) | 1 (3)
Polyuria (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Balanitis (Reproductive system and breast disorders) | 2 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (3)
Genital ulceration (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 1 (1)
Perineal ulceration (Reproductive system and breast disorders) | 1 (1)
Scrotal erythema (Reproductive system and breast disorders) | 1 (1)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (81)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (12)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 (31)
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Acne (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (6)
Eczema (Skin and subcutaneous tissue disorders) | 2 (3)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 4 (43)
Lichen planus (Skin and subcutaneous tissue disorders) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1)
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 6 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (11)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (3)
Rash (Skin and subcutaneous tissue disorders) | 11 (34)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (35)
Skin depigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 4 (5)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 2 (4)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (53)
Catheter removal (Surgical and medical procedures) | 1 (2)
Cautery to nose (Surgical and medical procedures) | 1 (1)
Central venous catheterisation (Surgical and medical procedures) | 1 (1)
Ear tube insertion (Surgical and medical procedures) | 1 (1)
Medical device removal (Surgical and medical procedures) | 4 (4)
Thrombectomy (Surgical and medical procedures) | 1 (1)
Flushing (Vascular disorders) | 4 (8)
Hot flush (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 3 (6)
Hypotension (Vascular disorders) | 2 (3)
Poor venous access (Vascular disorders) | 3 (6)
Thrombosis (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI cannot publish any data prior to multi-centre publication. If publication related to sub-sets of data it shall make reference to the relevant multi-centre publication. PI agrees to submit material to Sponsor for review at least 60 days prior to publication and incorporate all reasonable comments. During review, Sponsor may request that publication be delayed for up to 6 months from date of first submission to Sponsor in order for Sponsor to take steps to protect its proprietary information.